CLINICAL TRIAL: NCT04512976
Title: Exercise in Burn Survivors: Cooling Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Craig Crandall, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STU_2020_0334; 2R01GM068865-13A1 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-14 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Burn Injury
Keywords: skin graft; thermoregulation; burn survivor; 3rd degree burn injury; human
MeSH Terms: conditions — Burns | interventions — CCP110 protein, human

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized crossover design study. Burn survivors (20-40% burn surface area), burn survivors (>40% burn surface area), and non-burned individuals will each perform four bouts of 60-min of exercise trials with the following cooling strategies: A) a control trial, B) skin wetting only trial, C) fan only trial, and D) a combination of skin wetting with a fan trial. Subjects will perform these four bouts under one of the following environmental conditions (30 deg C and 38 deg C).
  A subject will only be required to perform exercise across all four cooling modalities for a given environmental temperature (i.e., four exercise bouts); each will not be required to perform exercise across all combinations of environmental temperatures and cooling modalities (i.e., 12 exercise bouts).
Masking Description: No masking is required as each subject will be exposed to each cooling modality (e.g., fan only, skin wetting, and a combination of a fan and skin wetting).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) (Experimental): Burn survivors with 20-40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (30°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
  Interventions: Other: Control (no cooling modalities); Other: Water Spray Only; Other: Fan Only; Other: Water Spray and Fan
- Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) (Experimental): Burn survivors with 20-40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (39°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
  Interventions: Other: Control (no cooling modalities); Other: Water Spray Only; Other: Fan Only; Other: Water Spray and Fan
- Non-Burned Individuals in Ambient Heat (30°C) (Experimental): Non-burned individuals will exercise for 60 minutes in ambient heat (30°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
  Interventions: Other: Control (no cooling modalities); Other: Water Spray Only; Other: Fan Only; Other: Water Spray and Fan
- Non-Burned Individuals in Ambient Heat (39°C) (Experimental): Non-burned individuals will exercise for 60 minutes in ambient heat (39°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
  Interventions: Other: Control (no cooling modalities); Other: Water Spray Only; Other: Fan Only; Other: Water Spray and Fan
- Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) (Experimental): Burn survivors with >40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (30°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
  Interventions: Other: Control (no cooling modalities); Other: Water Spray Only; Other: Fan Only; Other: Water Spray and Fan
- Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C) (Experimental): Burn survivors with >40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (39°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
  Interventions: Other: Control (no cooling modalities); Other: Water Spray Only; Other: Fan Only; Other: Water Spray and Fan

INTERVENTIONS:
Other: Control (no cooling modalities) — Subjects will exercise for 60 minutes in the indicated environmental condition while being exposed to no cooling modality.
Other: Water Spray Only — Subjects will exercise for 60 minutes in the indicated environmental condition while being exposed to the skin wetting modality.
  Skin wetting will be performed by spraying water onto the skin throughout the exercise bout.
Other: Fan Only — Subjects will exercise for 60 minutes in the indicated environmental condition while being exposed to the fan cooling modality.
  The fan will be a commercially available fan will be directed to the research subject throughout the exercise bout.
Other: Water Spray and Fan — Subjects will exercise for 60 minutes in the indicated environmental condition while being exposed to both the skin wetting and fan cooling modalities.
  The fan will be a commercially available fan will be directed to the research subject throughout the exercise bout.
  Skin wetting will be performed by spraying water onto the skin throughout the exercise bout.

SUMMARY:
This project will identify the efficacy of cooling modalities aimed to attenuate excessive elevations in skin and internal body temperatures during physical activity in well-healed burn survivors. The investigators will conduct a randomized crossover design study. Non-burned control subjects, subjects who experienced burns covering ~20% to 40% of their body surface area, and subject having burns >40% of their body surface area will be investigated. Subjects will exercise in heated environmental conditions while receiving the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of fan and skin wetting.

DETAILED DESCRIPTION:
Within the United States, 500,000+ individuals are enduring the long-term consequences of severe burn injuries covering 20% or more of their body surface area, with upwards to 11,000 individuals experiencing such an injury per year. These burn injuries can severely compromise body temperature regulation, owing to permanent impairments in the primary thermoeffectors necessary to dissipate heat, namely profoundly blunted skin blood flow and sweating responses in the injured skin. The investigators propose that this heat intolerance deters burn survivors from participating in physical activity, including activities of daily living, necessary to avoid the adverse cardiovascular and metabolic sequela of a sedentary lifestyle. Consistent with hypothesis, years after the injury burn survivors have a very low aerobic capacity; greater all-cause mortality rates; greater hospitalization days for circulatory diseases; and suffer from greater incidences of ischemic heart disease, heart failure, diabetes, and cerebrovascular disease (including stroke) relative to matched non-burned cohorts. The primary goal of this project is to identify modalities to attenuate excessive elevations in skin and core body temperatures during physical activity in well-healed burn survivors. The implementation of such modalities will eliminate heat intolerance as a barrier to participation in activities that are necessary to improve/maintain cardiovascular health in this vulnerable population. This project will investigate whether increased skin wetness, with and without accompanying fan use, will restore otherwise impaired evaporative cooling of well-healed burn survivors, with the extent of that improvement predicated on the environmental conditions and the percentage of body surface area burned.

ELIGIBILITY:
Inclusion Criteria (non-burned individuals):

* Healthy male and female subjects
* 18-65 years of age.
* Free of any underlying medical conditions

Exclusion Criteria (non-burned individuals):

* Any burn-related injuries resulting in at least one night of hospitalization.
* Heart disease or any other chronic medical condition requiring regular medical therapy including cancer, diabetes, and hypertension.
* Abnormalities detected on routine screening
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2.
* Pregnant individuals

Inclusion Criteria (burn survivors):

* Healthy male and female subjects
* 18-65 years of age.
* Free of any underlying medical conditions
* Having a burn injury covering 20-40% or >40% of the participant's body surface area; at least 50% of those burn injuries must be full thickness that required skin grafting.
* Participants must have been hospitalized due to the burn injury for a minimum of 15 days

Exclusion Criteria (burn survivors):

* Any burn-related injuries resulting in at least one night of hospitalization.
* Heart disease or any other chronic medical condition requiring regular medical therapy including cancer, diabetes, and hypertension.
* Abnormalities detected on routine screening
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2.
* Pregnant individuals
* Extensive unhealed injured skin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Exercise and Environmental Medincine - Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 70 subjects were enrolled in the study (signed the consent form). However, 5 of those subjects were screened out of the study during their consent visit due to elevated blood pressure (3), anxiety regarding the study procedures (1), and a body mass index higher than 35 (1).
Groups:
- Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C): Burn survivors with 20-40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (30°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (38°C): Burn survivors with 20-40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (38°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Non-Burned Individuals in Ambient Heat (30°C): Non-burned individuals will exercise for 60 minutes in ambient heat (30°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Non-Burned Individuals in Ambient Heat (38°C): Non-burned individuals will exercise for 60 minutes in ambient heat (38°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C): Burn survivors with >40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (30°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (38°C): Burn survivors with >40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (38°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
Period: Overall Study
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (38°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (38°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (38°C)
Started | 11 | 10 | 10 | 10 | 10 | 14
Completed | 11 | 10 | 10 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Unable to complete the exercise protocols in the study. | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: 65 subjects started this study, however, 3 were withdrawn prior to completing the study. Thus, our analyzed participant baseline information only includes 62 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (38°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (38°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (38°C) | Total
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 10 | 11 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 10 | 10 | 10 | 11 | 62
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 5 | 5 | 5 | 31
  Male | 5 | 5 | 5 | 5 | 5 | 6 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 7 | 9 | 8 | 8 | 7 | 47
  African American/Black | 3 | 3 | 1 | 2 | 1 | 3 | 13
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Non-Hispanic | 10 | 9 | 8 | 9 | 9 | 10 | 55
  Hispanic | 1 | 1 | 2 | 1 | 1 | 1 | 7
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.48 (3.86) | 25.76 (3.64) | 23.57 (1.89) | 23.85 (1.97) | 27.77 (3.45) | 27.12 (2.62) | 25 (3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Temperature (°C) During Control Intervention
Description: The subject's core body temperature will be measured from gastrointestinal temperature via an ingestible telemetric pill.
Time Frame: At 0 minutes and 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Non-Burned Individuals in Ambient Heat (30°C) | Non-Burned Individuals in Ambient Heat (39°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 11
°C | .578 (.270) | .920 (.432) | .622 (.205) | .885 (.404) | .863 (.449) | 1.29 (.580)

2. Primary Outcome: Change in Core Temperature (°C) During Fan Intervention
Description: as for outcome 1
Time Frame: At 0 minutes and 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Groups:
- Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C): Burn survivors with 20-40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (39°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Non-Burned Individuals in Ambient Heat (39°C): Non-burned individuals will exercise for 60 minutes in ambient heat (39°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C): Burn survivors with >40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (39°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 11
°C | .537 (.195) | .996 (.654) | .728 (.318) | .891 (.267) | .838 (.463) | 1.135 (.565)

3. Primary Outcome: Change in Core Temperature (°C) During Water-Spray Intervention
Description: as for outcome 1
Time Frame: At 0 minutes and 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 11
°C | .511 (.224) | .922 (.289) | .726 (.222) | .792 (.372) | .787 (.294) | .940 (.488)

4. Primary Outcome: Change in Core Temperature (°C) During Water-Spray and Fan Intervention
Description: as for outcome 1
Time Frame: At 0 minutes and 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 11
°C | .630 (.260) | .869 (.354) | .604 (.285) | .928 (.347) | .858 (.331) | .928 (.453)

5. Secondary Outcome: Skin Temperature (°C) Following Control Intervention
Description: The subject's skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin.
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Non-Burned Individuals in Ambient Heat (30°C) | Non-Burned Individuals in Ambient Heat (39°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10 | 9
°C | 33.204 (1.737) | 37.149 (1.606) | 30.978 (1.096) | 35.863 (2.339) | 34.092 (1.685) | 37.146 (1.106)

6. Secondary Outcome: Skin Temperature (°C) Following Fan Intervention
Description: as for outcome 5
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 8 | 10 | 10 | 10 | 9
°C | 32.787 (1.862) | 37.660 (1.435) | 30.396 (1.243) | 33.911 (2.005) | 32.819 (1.237) | 37.146 (1.106)

7. Secondary Outcome: Skin Temperature (°C) Following Water-Spray Intervention
Description: as for outcome 5
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
°C | 29.114 (2.665) | 34.332 (2.535) | 29.110 (2.101) | 32.879 (1.165) | 28.65 (3.559) | 33.549 (2.839)

8. Secondary Outcome: Skin Temperature (°C) Following Water-Spray and Fan Intervention
Description: as for outcome 5
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
°C | 28.727 (3.565) | 34.406 (3.914) | 27.276 (2.647) | 32.659 (2.574) | 26.958 (3.039) | 34.661 (3.242)

9. Secondary Outcome: Heart Rate Following Control Intervention
Description: The subject's heart rate will be measured from ECG electrodes attached to the participant.
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Non-Burned Individuals in Ambient Heat (30°C) | Non-Burned Individuals in Ambient Heat (39°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10 | 11
beats per minute | 113 (17) | 128 (24) | 110 (14) | 118 (9) | 117 (21) | 142 (27)

10. Secondary Outcome: Heart Rate Following Fan Intervention
Description: The subject's heart rate will be measured from ECG electrodes attached to the participant.
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10 | 11
beats per minute | 114 (18) | 133 (29) | 106 (13) | 125 (13) | 113 (22) | 136 (25)

11. Secondary Outcome: Heart Rate Following Water-Spray Intervention
Description: The subject's heart rate will be measured from ECG electrodes attached to the participant.
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 11
°C | 113 (16) | 132 (24) | 112 (14) | 118 (11) | 113 (21) | 130 (18)

12. Secondary Outcome: Heart Rate Following Water-Spray and Fan Intervention
Description: The subject's heart rate will be measured from ECG electrodes attached to the participant.
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 9 | 11
°C | 112 (15) | 129 (24) | 107 (12) | 120 (17) | 112 (19) | 128 (25)

13. Secondary Outcome: Mean Arterial Blood Pressure Following Control Intervention
Description: The subject's mean arterial blood pressure will be measured using a standard arm blood pressure cuff.
  Mean Arterial Pressure (MAP) is a common physiological measure calculated by adding the diastolic blood pressure value to one third of the difference between the systolic (SBP) and diastolic (DBP) blood pressure values.
  MAP = DBP + 1/3(SBP - DBP)
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Non-Burned Individuals in Ambient Heat (30°C) | Non-Burned Individuals in Ambient Heat (39°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 9 | 8 | 10 | 10 | 10 | 10
mmHg | 89 (9) | 86 (10) | 86 (12) | 83 (7) | 100 (15) | 97 (11)

14. Secondary Outcome: Mean Arterial Blood Pressure Following Fan Intervention
Description: as for outcome 13
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 8 | 7 | 10 | 10 | 10 | 11
mm Hg | 94 (10) | 94 (12) | 89 (14) | 86 (10) | 97 (14) | 89 (20)

15. Secondary Outcome: Mean Arterial Blood Pressure Following Water-Spray Intervention
Description: as for outcome 13
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 9 | 8 | 9 | 9 | 9 | 10
mm Hg | 91 (14) | 96 (10) | 82 (9) | 82 (9) | 104 (19) | 96 (12)

16. Secondary Outcome: Mean Arterial Blood Pressure Following Water-Spray and Fan Intervention
Description: as for outcome 13
Time Frame: At 60 minutes into the intervention.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (39°C) | Experimental: Non-Burned Individuals in Ambient Heat (30°C) | Experimental: Non-Burned Individuals in Ambient Heat (39°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Experimental: Burn Survivors (>40% Burn Surface Area) in Ambient Heat (39°C)
Number analyzed (Participants) | 10 | 9 | 10 | 9 | 9 | 10
mm Hg | 94 (15) | 88 (6) | 90 (12) | 84 (9) | 95 (13) | 92 (16)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the 4 trial protocol for each subject.
Groups:
- Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (38°C): Burn survivors with 20-40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (38°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Non-Burned Individuals in Ambient Heat (38°C): Non-burned individuals will exercise for 60 minutes in ambient heat (38°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
- Burn Survivors (>40% Burn Surface Area) in Ambient Heat (38°C): Burn survivors with >40% BSA (burn surface area) will exercise for 60 minutes in ambient heat (38°C) while being exposed to each of the following cooling modalities: no cooling, fan only, skin wetting only, and a combination of a fan and skin wetting.
Arm/Group | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (20-40% Burn Surface Area) in Ambient Heat (38°C) | Non-Burned Individuals in Ambient Heat (30°C) | Non-Burned Individuals in Ambient Heat (38°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (30°C) | Burn Survivors (>40% Burn Surface Area) in Ambient Heat (38°C)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT04512976/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT04512976/ICF_001.pdf